CLINICAL TRIAL: NCT06657703
Title: A Phase Ia Single Center, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single Doses of HC022 in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single Doses of HC022 in Healthy Subjects.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HC Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC022-I-001
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- HC022 5mg SC (Experimental): Participants will receive single subcutaneous (SC) dose of 5 mg HC022 or matching placebo on Day 1.
  Interventions: Drug: HC022; Drug: Placebo
- HC022 50mg SC (Experimental): Participants will receive single subcutaneous (SC) dose of 50 mg HC022 or matching placebo on Day 1.
  Interventions: Drug: HC022; Drug: Placebo
- HC022 150mg SC (Experimental): Participants will receive single subcutaneous (SC) dose of 150 mg HC022 or matching placebo on Day 1.
  Interventions: Drug: HC022; Drug: Placebo
- HC022 450mg SC (Experimental): Participants will receive single subcutaneous (SC) dose of 450 mg HC022 or matching placebo on Day 1.
  Interventions: Drug: HC022; Drug: Placebo
- HC022 900mg SC (Experimental): Participants will receive single subcutaneous (SC) dose of 900 mg HC022 or matching placebo on Day 1.
  Interventions: Drug: HC022; Drug: Placebo

INTERVENTIONS:
Drug: HC022 — Administered as specified in the treatment arm
Drug: Placebo — Administered as specified in the treatment arm

SUMMARY:
The primary objective of this phase Ia study is to evaluate the safety and tolerability of single-ascending, subcutaneous (SC) doses of HC022 in healthy subjects. Secondary objectives of study are as follows: To estimate the PK parameters of single-ascending SC doses of HC022 in healthy subjects；To evaluate the immunogenicity of HC022 administered to healthy subjects.

DETAILED DESCRIPTION:
This is a first-in-human study of HC022 to assess safety, tolerability, and pharmacokinetic (PK) and pharmacodynamic (PD) effects of single HC022 doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and comply with study requirements;
2. Aged 18 to 55 years old, inclusive, male or female;
3. 3.A body weigh ≥ 50 kg for male , and a body weigh ≥ 45 kg for female, and must have a body mass index between 19 and 28 kilogram per square meter (kg/m2)；
4. Be in good health as based on medical history, physical examination, vital signs, laboratory tests, chest radiographs, abdominal ultrasound and 12-lead ECG；
5. All women of childbearing potential and all men must practice highly effective contraception during the study and for 6 months (for female) or 3 months (for male) after their dose of study treatment；

Exclusion Criteria:

1. Have participated in other clinical trials within 3 months, or within the 5 half lives of the investigational drug prior to screening, whichever is longer;
2. History of or positive test results at screening for the following: for human immunodeficiency virus (HIV), hepatitis C virus antibody (HCV Ab), hepatitis B virus (defined as positive for HBsAg or HBcAb or HBeAg)；
3. History of or current diagnosis of active tuberculosis (TB), or untreated latent TB infection (LTBI) at screening；
4. History of severe herpes infection or zoster viral infection；
5. Serious infection, serious injuries, or major surgical procedures within 6 months prior to Screening；
6. History of alcohol or substance abuse, a positive urine drug or alcohol test at Day -1；
7. History of severe allergic or anaphylactic reactions or history of allergic reactions likely to be exacerbated by any component of the study drug；
8. Any disease or conditons that are not suitable for participation in this study as determined by the Investigator；

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 20 weeks

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 Extrapolated to Infinity (AUCinf) of HC022 | Up to 20 weeks
Maximum Observed Concentration (Cmax) of HC022 | Up to 20 weeks
Time to Reach Maximum Observed Concentration (Tmax) of HC022 | Up to 20 weeks
Terminal Elimination Half-Life (t1/2) of HC022 | Up to 20 weeks
Apparent Clearance (CL/F) of HC022 | Up to 20 weeks
Apparent Volume of Distribution (Vz/F) of HC022 | Up to 20 weeks
Number of Participants Who Develop Serum Anti-HC022 Antibodies | Up to 20 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing
  - The Clinical Pharmacology Research Center of PUMCH, Beijing